CLINICAL TRIAL: NCT00002684
Title: Phase II Trial of Paclitaxel, Cisplatin and Ifosfamide in Patients With Advanced Urothelial Tumors
Brief Title: Combination Chemotherapy in Patients With Advanced Urinary Tract Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Purpose: Treatment
Other Study IDs: 95-031; CDR0000064373 (Registry Identifier: PDQ (Physician Data Query)); NCI-V95-0743
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-07

CONDITIONS: Bladder Cancer; Urethral Cancer
Keywords: stage III bladder cancer; recurrent bladder cancer; stage IV bladder cancer; squamous cell carcinoma of the bladder; adenocarcinoma of the bladder; recurrent urethral cancer; distal urethral cancer; proximal urethral cancer; urethral cancer associated with invasive bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urethral Neoplasms | interventions — Cisplatin; Ifosfamide; Paclitaxel

INTERVENTIONS:
Drug: cisplatin
Drug: ifosfamide
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cisplatin, ifosfamide, and paclitaxel, use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug and giving drugs in different ways may kill more tumor cells.

PURPOSE: This phase II trial is studying how well combination chemotherapy works in treating patients with metastatic urinary tract cancer that cannot be treated with surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of cisplatin, ifosfamide, and paclitaxel in patients with unresectable or metastatic urothelial cancer (nontransitional cell histologies).

OUTLINE: Patients receive paclitaxel IV over 3 hours and cisplatin IV over 1 hour on day 1 and ifosfamide IV over 1 hour on days 1-3. Filgrastim (G-CSF) is administered subcutaneously daily beginning on day 6 and continuing through day 17 or until blood counts recover. Treatment continues every 3 weeks for a maximum of 6 courses in the absence of stable or progressive disease after completion of course 2 or complete response after completion of course 4.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven unresectable or metastatic urothelial cancer

  * No transitional cell histologies
* Bidimensionally measurable disease

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Hematopoietic:

* WBC at least 3,500/mm^3
* Platelet count greater than 150,000/mm^3

Hepatic:

* Bilirubin less than 2.0 mg/dL

Renal:

* Creatinine less than 1.5 mg/dL OR
* Creatinine clearance greater than 55 mL/min

Cardiovascular:

* No New York Heart Association class III or IV heart disease

Other:

* No other concurrent malignancy except basal cell skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior systemic chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* At least 3 weeks since prior radiotherapy

Surgery

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 1995-05; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Dean F. Bajorin, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States